CLINICAL TRIAL: NCT00640237
Title: Vitamin D Deficiency in the Elder Patients of General Departments and Its Treatment During the Hospitalization
Brief Title: Interventional Trial of Vitamin D Deficiency in the Patients of General Departments
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Professor Sofia Ish-Shalom, The Chief of Unite for Bone Metabolism of Rambam Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VD-1.CTIL
Record Dates: First submitted 2008-03-16; First posted 2008-03-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamine D State
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Calcifediol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Arm 1 - the patients will receive two large doses of vitamin D.
  Interventions: Dietary Supplement: Alpha-D3
- 2 (No Intervention): Arm 2 - the patients vitamin D status will be checked during the hospitalization and they will receive the recommendation to treat the vitamin D deficiency in the out-patient department.

INTERVENTIONS:
Dietary Supplement: Alpha-D3 — We will use the vitamin alpha-D3 drops of CTS pharmaceutical firm , that contains 5000 IU in ml. Every patient in the interventional group will receive two dose of 100000 IU (20 ml)vitamin alpha-D3 within a month period.
  Other Names: 25(OH)-D3
  Arms: 1

SUMMARY:
The purpose of the study is to examine the vitamin D state of elder patients in therapeutic departments and to compere the treatment during the hospitalization with the out-patient treatment.

DETAILED DESCRIPTION:
Today vitamin D is thought to be one of the most important vitamins in the human body. It's made in the skin during the sun expose, so it must be sufficient in so sunny countries as Israel. Although many old people in our country suffer from vitamin d deficiency which bring them to recurrent falls, osteoporotic fractures and physical disability. This problem is still underestimated by health authorities in different countries.

In this study we will examine the vitamin D state of the therapeutic patient older than 65 year including their physical self-estimation, muscle strength measurement and gait-and-balance tests. Then, according to the resent studies, we will treat the patients in the interventional group with two large doses of vitamin D during a month. After that we will compere their health and physical state with the patients treated in the out-hospital department.

So we will try to find a useful approach to treat the vitamin D deficiency during the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* the patient was admitted to a general department of Rambam Medical Center for any reason from March to May 2008
* the patient is 65 years old or older
* the patient is in a good health, based on medical history, physical examination and laboratory screening evaluation.

Exclusion Criteria:

* renal failure with creatinine level more then 1.3 mg/dL or nephritic syndrome.
* liver disease with transaminase rise three times from normal level.
* nephrolithiasis in the last fife years.
* primary hyperparathyroidism, hypoparathyroidism or pseudohypoparathyroidism.
* advanced cancer.
* chronic diarrhea or malabsorption.
* granulomatous disease (sarcoidosis, tuberculosis, lymphoma).
* patients, who are receiving barbiturates, rifampin, anticonvulsants.
* patients, who are receiving digitalis.
* patients, who are receiving glucocorticoids for more than two weeks during the study.
* advanced dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-07 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
vitamin D status | two month

SECONDARY OUTCOMES:
physical performance, health conditions, arm strength, gait and balance state. | two month

CONTACTS AND LOCATIONS:
Overall Officials: Ish-Shalom Sofia, Professor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel